CLINICAL TRIAL: NCT03079661
Title: Impact of Air Quality on Exacerbations of COPD in the Somme
Acronym: PolluBPCO
Status: Terminated | Type: Observational
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-42
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Acute Exacerbation Copd
Keywords: pollution; ozone; Copd; particles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All COPD patients with a diagnosis of acute exacerbation in emergency room in University Hospital of Amiens-Picardie between 01/01/2017 and 31/12/2017. The investigator will collect for each patient the home address and the work address. The duration of 1 year was chosen to take into account seasonal variations. In parallel, a daily report of the rate of ozone, particles (PM2.5 and PM10), dioxide nitrogen but also odours and pollens will be done by ATMO Picardie.

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients with a diagnosis of acute exacerbation of COPD in the emergency room. The definition of COPD and acute exacerbation are the official definition of the Société de Pneumologie en Langue Française.

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The primary endpoint is the number of exacerbations of COPD corresponding to the variable of interest to be explained. The other variables are the explanatory variables (air quality data PM2.5, PM10, NO2, O3 as well as pollen data, seasonal variations, influenza epidemic and olfactory nuisance). The final diagnosis will also be collected.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
exacerbation rate : variable to be explicated with explicative variable : ozone, particles, dioxide nitrogen, but also pollens corresponding to each patient home address for period of exacerbation | 1 day
  exacerbation rate : variable to be explicated with explicative variable : ozone, particles, dioxide nitrogen, but also pollens corresponding to each patient home address for period of exacerbation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Derived] Basille D, Soriot L, Weppe F, Desmettres P, Henriques P, Benoit N, Devaux S, Diouf M, Jounieaux V, Andrejak C. Association between acute exacerbation of chronic obstructive pulmonary disease and short-term exposure to ambient air pollutants in France. Environ Health. 2024 Nov 29;23(1):107. doi: 10.1186/s12940-024-01146-3. PMID 39614356